CLINICAL TRIAL: NCT03065634
Title: Return to Work and Living Healthy After Head and Neck Cancer
Acronym: RELIANCE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient recruitment rate
Sponsor: University of Leipzig (Other)
Collaborators: Universitätsklinikum Leipzig (Other); Jena University Hospital (Other); Klinikum St. Georg gGmbH (Other); Stadtisches Klinikum Dresden (Other); German Cancer Aid (Other)
Responsible Party: Principal Investigator, Anja Mehnert, Prof. Dr., University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 93000-133
Record Dates: First submitted 2017-02-17; First posted 2017-02-28 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Return to Work

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manualized RELIANCE intervention (Experimental): Return to work and living healthy after head and neck cancer (RELIANCE) is a 2-months group intervention for head and neck cancer patients delivered by a trained psychotherapist and a peer in eight sessions.
  Interventions: Behavioral: Return to work and living healthy after head and neck cancer
- Non-manualized socio-legal counseling (Active Comparator): two socio-legal counseling sessions delivered by a social worker
  Interventions: Behavioral: socio-legal counseling

INTERVENTIONS:
Behavioral: Return to work and living healthy after head and neck cancer — Return to work and living healthy after head and neck cancer (RELIANCE) is a 2-months group intervention for head and neck cancer patients delivered by a trained psychotherapist and a peer in eight sessions. The individual sessions aim to improve work ability, quality of life and psychological well-being
  Arms: Manualized RELIANCE intervention
Behavioral: socio-legal counseling — Non-manualized socio-legal counseling
  two socio-legal counseling sessions delivered by a social worker
  Arms: Non-manualized socio-legal counseling

SUMMARY:
Based on a randomized controlled trial, the manualized group intervention Return to work and living healthy after head and neck cancer (RELIANCE) for head and neck cancer survivors will be tested against a non-manualized control intervention (social counseling) in order to evaluate the efficacy of the RELIANCE intervention compared to the control condition. The study design includes two phases, the initial study phase (pilot study) and the intervention study (RCT). The aim of the pilot study is to implement and ensure the necessary standardized procedures for the implementation of patient recruitment and interventions. In the randomized controlled trial, potential participants are assigned to the intervention group or to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of laryngea, hypopharyngeal, oropharyngeal, tonsil or base of the tongue cancer within the last six months
* Curative treatment
* Completion of primary and follow-up Treatment
* Fluency in German
* Written informed and voluntary consent
* Psychological distress (Distress Thermometer score > 4)
* Self-perceived prognosis of employment (SPE score ≥ 1)

Exclusion Criteria:

* Alcohol dependency with physical withdrawal symptoms (CAGE score ≥ 3 and current use of alcohol)
* Acute suicidal tendencies
* Receiving old-age pension or will receive old-age pension within the next 12 months
* Cognitive impairment indicated in the medical records or by the attending doctor
* Being in psychotherapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 39 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Work ability | directly after intervention and at six months follow-up
  Work-Ability-Index, short version (WAI)
Pattern of work-related coping behaviour | directly after intervention and at six months follow-up
  Pattern of work-related coping behaviour, short Version (AVEM-44)

SECONDARY OUTCOMES:
Cancer-specific health-related quality of Life (global, functioning, symptom burden) | directly after intervention and at six months follow-up
  Quality of Life Core Questionnaire of the European Organisation for Research and Treatment of Cancer (EORTC-QLQ-C30)
Quality of life and symptoms specific to head and neck cancer | directly after intervention and at six months follow-up
  Head and Neck Module of the European Organisation for Research and Treatment of Cancer (EORTC-H&N35)
anxiety, depression and psychological distress in patients with somatic diseases | directly after intervention and at six months follow-up
  Hospital Anxiety and Depression Scale (HADS)
health behavior and health related attitudes and knowledge about specific diseases | directly after intervention and at six months follow-up
  questionnaire measuring health behavior and health related attitudes and knowledge about specific diseases (FEG)
general self-efficacy expectation | directly after intervention and at six months follow-up
  general self-efficacy expectation (ASKU)

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Leipzig, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://medpsy.uniklinikum-leipzig.de/medpsych.site,postext,projekte-psychoonkologie-aktuell,a_id,8222.html